CLINICAL TRIAL: NCT05562830
Title: A Phase 1/2 Open-Label Rolling-Arm Umbrella Platform Study of Investigational Agents With or Without Pembrolizumab in Participants With PD-1/L1 Refractory Locally Advanced or Metastatic Urothelial Carcinoma (KEYMAKER-U04): Substudy 04A
Brief Title: A Substudy of Investigational Agents in Programmed Cell Death-1/Ligand 1 (PD-1/L1) Refractory Locally Advanced or Metastatic Urothelial Carcinoma (mUC) (MK-3475-04A)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-04A; MK-3475-04A (Other: MSD); 2023-506384-34-00 (Registry Identifier: EU CT); U1111-1293-7548 (Registry Identifier: UTN); 2020-004544-28 (EudraCT Number)
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Zilovertamab vedotin (Experimental): Participants will receive zilovertamab vedotin 2mg/kg administered on Day 1 and Day 8 of each 3 week cycle (Q3W) until documented disease progression or any other discontinuation criterion is met.
  Interventions: Biological: Zilovertamab vedotin
- Arm B: Pembrolizumab and MK-3120 (Experimental): Participants will receive MK-3120 up to 5mg/kg administered on Day 1, Day 15 and Day 29 of each 6 week cycle until documented disease progression or any other discontinuation criterion is met and 400mg pembrolizumab on Day 1 of each 6 week cycle for up to 17 cycles (up to ~2 years).
  Interventions: Biological: Pembrolizumab; Biological: MK-3120

INTERVENTIONS:
Biological: Zilovertamab vedotin — Administered via intravenous (IV) infusion on day 1 and day 8 of Q3W cycles
  Other Names: MK-2140; VLS-101
  Arms: Arm A: Zilovertamab vedotin
Biological: Pembrolizumab — Administered via IV infusion on Day 1 of each 6 week cycle.
  Other Names: MK-3475; KEYTRUDA®
  Arms: Arm B: Pembrolizumab and MK-3120
Biological: MK-3120 — Administered as an IV infusion on Day 1, Day 15, and Day 29 of each 6 week cycle.
  Arms: Arm B: Pembrolizumab and MK-3120

SUMMARY:
This substudy is part of an umbrella platform study which is designed to evaluate investigational agents with or without pembrolizumab in participants with urothelial carcinoma who are in need of new treatment options. Substudy 04A will enroll participants with locally advanced or mUC whose disease is resistant to treatment with programmed cell death-1/ligand 1 (PD-1/L1) inhibitors. The protocol infrastructure will enable the rolling assignment of investigational treatments.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion and exclusion criteria include but are not limited to the following:

* Histologically or cytologically confirmed diagnosis of locally advanced/unresectable or mUC of the renal pelvis, ureter (upper urinary tract), bladder, or urethra.
* Arm A: PD-1/L1 refractory locally advanced or mUC as evidenced by: EITHER disease progression while on treatment or after treatment with an anti-PD-1/L1 monoclonal antibody (mAb) for locally advanced/unresectable or mUC administered either as monotherapy, or in combination with other checkpoint inhibitors or other therapies OR disease recurrence while on treatment or after treatment with an anti-PD-1/L1 mAb for muscle-invasive urothelial carcinoma (MIUC) administered as monotherapy.
* Arm A: Participants must provide an archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion demonstrating UC, not previously irradiated, and adequate for biomarker evaluation.
* Arm B: PD-1/L1 refractory locally advanced or mUC as evidenced by: EITHER disease progression after treatment with an anti-PD-1/L1 mAb for locally advanced/unresectable or mUC administered either as monotherapy, or in combination with other checkpoint inhibitors or other therapies; OR disease recurrence after treatment with an anti-PD-1/L1 mAb for MIUC administered as monotherapy or in combination with other checkpoint therapies >12 months after last dose of treatment with an anti-PD-1/L1 mAb.
* Arm B: Participants must provide an archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion from a metastatic site or from a primary tumor that has become locally advanced and not previously irradiated.

Exclusion Criteria:

* Known additional nonurothelial malignancy that is progressing or has required active treatment within 3 years prior to study randomization/allocation.
* Received prior systemic anticancer therapy including investigational agents within 4 weeks before randomization/allocation.
* Active infection requiring systemic therapy.
* Received a live or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines are allowed.
* Known history of human immunodeficiency virus (HIV).
* Known history of hepatitis B or known hepatitis C virus infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-11-16 (Actual); Primary Completion 2028-06-20 (Estimated); Study Completion 2028-06-20 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Who Experienced At Least One Adverse Event (AE) | Up to approximately 5 years
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment.
Percentage of Participants Who Discontinued Study Treatment Due to an AE | Up to approximately 5 years
  An AE is defined as any unfavorable and unintended sign, symptom, disease, or worsening of preexisting condition temporally associated with study treatment and irrespective of causality to study treatment
Arm A: Objective Response Rate (ORR) as Assessed by Blinded Independent Central Review (BICR) | Up to approximately 2 years
  ORR is defined as the percentage of participants who achieve a Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria In Solid Tumors Version 1.1 (RECIST 1.1). The percentage of participants who experience CR or PR as assessed by Blinded Independent Central Review (BICR) will be presented.
Arm B: ORR as Assessed by Investigator | Up to approximately 2 years
  ORR is defined as the percentage of participants who achieve a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1. The percentage of participants who experience CR or PR as assessed by the investigator will be presented.

SECONDARY OUTCOMES:
Arm A: Duration of Response (DOR) as Assessed by BICR | Up to approximately 2 years
  For participants who demonstrate confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by Blinded Independent Central Review (BICR) will be presented.
Arm B: DOR as Assessed by Investigator | Up to approximately 2 years
  For participants who demonstrate confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until PD or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by the investigator will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (26):
- United States (9):
  - University of California, Irvine (UCI) Health - UC Irvine Medical Center ( Site 1045), Orange, California
  - University of California San Francisco ( Site 1044), San Francisco, California
  - Anschutz Cancer Pavilion ( Site 1017), Aurora, Colorado
  - University of Chicago Medical Center ( Site 1037), Chicago, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center ( Site 1011), Indianapolis, Indiana
  - Siteman Cancer Center ( Site 1038), St Louis, Missouri
  - Cleveland Clinic-Taussig Cancer Center ( Site 1036), Cleveland, Ohio
  - UPMC Hillman Cancer Center ( Site 1014), Pittsburgh, Pennsylvania
  - Huntsman Cancer Institute ( Site 1041), Salt Lake City, Utah
- Royal Brisbane and Women's Hospital-Medical Oncology Clinical Trials Unit, Cancer Care Services ( Site 1952), Brisbane, Queensland, Australia
- Chile (2):
  - FALP-UIDO ( Site 1151), Santiago, Region M. de Santiago
  - Bradford Hill ( Site 1155), Santiago, Region M. de Santiago
- Rigshospitalet-Dept. of Oncology ( Site 1701), Copenhagen, Capital Region, Denmark
- Israel (3):
  - Rambam Health Care Campus-Oncology ( Site 1501), Haifa
  - Rabin Medical Center-Oncology ( Site 1504), Petah Tikva
  - Sheba Medical Center-ONCOLOGY ( Site 1503), Ramat Gan
- Italy (2):
  - Fondazione IRCCS Istituto Nazionale dei Tumori-Struttura Complessa Oncologia Medica 1 ( Site 1408), Milan, Lombardy
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale-S.C. Sperimentazioni Cliniche ( Site 1406), Napoli
- Nederlands Kanker Instituut - Antoni van Leeuwenhoek (NKI-AVL)-medical oncology ( Site 1302), Amsterdam, North Holland, Netherlands
- South Korea (3):
  - Severance Hospital, Yonsei University Health System ( Site 1903), Seoul
  - Asan Medical Center ( Site 1901), Seoul
  - Samsung Medical Center ( Site 1902), Seoul
- Spain (2):
  - Hospital Universitari Vall d'Hebron ( Site 1767), Barcelona, Catalonia
  - Hospital Clinico San Carlos ( Site 1765), Madrid
- United Kingdom (2):
  - St Bartholomew's Hospital ( Site 1206), London, London, City of
  - ROYAL MARSDEN HOSPITAL (CHELSEA) ( Site 1201), London, London, City of

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com
- See also: Protocol Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26276&tenant=MT_MSD_9011